CLINICAL TRIAL: NCT06598592
Title: Video Emergency Calls of Bystanders - a Simulation Study
Brief Title: Video Emergency Calls of Bystanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Principle Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Video-Emergency-Call
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-09

CONDITIONS: Audio-Emergency Call; Video-Emergency Call

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Audio Emergency Call (Sham Comparator): An Emergency Call will be performed
  Interventions: Other: Audio-Emergency Call
- Video-Emergency Call (Active Comparator): Video-Emergency Call
  Interventions: Other: Video-Emergency

INTERVENTIONS:
Other: Video-Emergency — Video Emergency Call using a webbased platform
  Arms: Video-Emergency Call
Other: Audio-Emergency Call — Audio Emergency Call
  Arms: Audio Emergency Call

SUMMARY:
Emergency center dispatchers often face the challenge that emergency calls typically provide only verbal information. However, many first responders use smartphones, which could enable the option for video calls during emergencies. Leveraging this technology could offer control center staff additional insights, potentially transforming the way they manage emergency situations. Despite this, the impact of video emergency calls on call duration and user experience remains largely unexplored.

In this project, 20 control center employees will undergo a one-hour training session on a video emergency call system. After the training, each dispatcher will handle four simulated emergency calls-two via audio and two via video. To facilitate this, 80 first responders will be recruited from public spaces, such as shopping centers. These responders will face simulated emergencies, including epileptic seizures, shortness of breath, forehead lacerations, or injuries to the upper extremities with minor bleeding. Professional medical actors will simulate the emergencies, and the responders will be tasked with making either an audio or video emergency call.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* User of a smartphone
* German Language

Exclusion Criteria:

* EMS personnel

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Duration of the Emergency Call | Up to 10 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No